CLINICAL TRIAL: NCT02818283
Title: Soy Modulation of Immune Activation, LDL- Levels, and Lowering Inflammation by Pretzel Isoflavone Dietary Intervention
Acronym: SMALLLIPIDS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment and funding
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Nicholas Funderburg, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015H0375
Record Dates: First submitted 2016-06-16; First posted 2016-06-29 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection; Hypercholesterolemia
Keywords: Human Immunodeficiency Virus; hypercholesterolemia; pretzels; nutritional study; dietary soy; antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Soy Pretzel-Short Feasibility (Experimental): 6 week intervention involving daily consumption of soy pretzel (two packets, 5 oz./packet) for 28 days. Participants will follow a legume-free diet which restricts the consumption of legume foods (soy, beans, peas, peanuts, and lentils) during the study period. This arm will precede the longer 28 week study
  Interventions: Dietary Supplement: Soy Pretzel
- Soy Pretzel (Active Comparator): 28 week intervention involving daily consumption of soy pretzel (two packets, 5 oz./packet) for 12 weeks. Participants will follow a legume-free diet which restricts the consumption of legume foods (soy, beans, peas, peanuts, and lentils) during the study period. Participants will be randomized to start with soy pretzel or wheat pretzel arm and crossover to the other pretzel at week 14.
  Interventions: Dietary Supplement: Soy Pretzel
- Wheat Pretzel (Placebo Comparator): 28 week intervention involving daily consumption of wheat pretzel (two packets, 5 oz./packet) for 12 weeks. Participants will follow a legume-free diet which restricts the consumption of legume foods (soy, beans, peas, peanuts, and lentils) during the study period. Participants will be randomized to start with soy pretzel or wheat pretzel arm and crossover to the other pretzel at week 14.
  Interventions: Other: Wheat Pretzel

INTERVENTIONS:
Dietary Supplement: Soy Pretzel — Each packet (5oz.) of soy pretzel contains high gluten wheat flour, soy flour, soymilk, vegetable shortening, sugar, yeast, salt, and ascorbic acid. Each packet provides ~280 calories (16% fat, 54% total carbohydrates, and 30% protein).
  Arms: Soy Pretzel; Soy Pretzel-Short Feasibility
Other: Wheat Pretzel — Each packet (5oz.) of wheat pretzel contains high gluten wheat flour, vital wheat gluten, shortening, sugar, yeast, salt, and ascorbic acid. Each packet provides ~290 calories (16% fat, 54% total carbohydrates, and 30% protein).
  Arms: Wheat Pretzel

SUMMARY:
Combination antiretroviral therapy (ART, HIV medications) dramatically increases the expected lifespan of HIV (Human Immunodeficiency Virus)infected patients; yet, the risks for cardiovascular disease (CVD), such as heart attacks and stroke, are increased in this population. This increased risk may be linked to persistent inflammation and activation of the immune system. Although the relationship between cardiovascular disease and HIV-infected individuals who are taking HIV medications is not well understood, the team of researchers involved in this study observed that a diet rich in soy, at levels recommended by the FDA (Federal Drug Administration), improved cholesterol levels and inflammation in individuals not infected with HIV. From this study, the researchers hope to gain understanding on how dietary soy will impact HIV-infected individuals who are taking HIV medications. Two pretzels with and without soy developed at OSU (Ohio State University) in the Department of Food Science and Technology and used in previous clinical trials will be used to investigate how the pretzel snacks will affect your cardiovascular disease risk, immunity, and how your body breaks down naturally occurring chemicals from soy.

DETAILED DESCRIPTION:
This study will significantly advance our knowledge of how dietary soy impacts lipid levels and composition, metabolic parameters and inflammation in HIV+ patients treated with anti-retroviral therapy (ART). HIV+ persons are at increased risk for CVD, and both HIV and ART are associated with metabolic perturbations (including lipid disturbances) and chronic inflammation. There is growing recognition that correcting these perturbations may improve life expectancy. Two clinical trials, first a short-term single armed study, followed by a two armed, placebo controlled, crossover clinical trial, will be used to address the feasibility of a soy-based, functional food intervention and the impact of that intervention on metabolic and immunomodulatory parameters. Daily pretzel dosing of two packets was determined from prior clinical trials with soy bread in patients with prostate cancer. The use of a food-based delivery vehicle has many advantages compared to using a dietary supplement as it provides a strategy to deliver a complexity of bioactive compounds found only in whole food ingredients. We hypothesize that the soy pretzel formulation will be well tolerated with excellent adherence (>95%) among ART-treated HIV+ patients with moderate hypercholesterolemia. The short-term dose confirmation study (n=20) will be a 6 week study using a single intervention and single dose of soy pretzels to determine Grade 1 and 2 toxicities, compliance, and tolerability of soy pretzels in ART-treated HIV+ patients with moderate hypercholesterolemia. Once, we have confirmed the short-term feasibility of soy pretzels, a subsequent longer-term study will involve a 28 week randomized, placebo-controlled, crossover trial (n=80) with soy and wheat (placebo) pretzels. Overall, the short-term dose confirmation study will provide the necessary clinical data required to move this intervention forward to the long-term placebo controlled trial. Both studies will provide us with valuable biologic material to assess changes in cardiovascular and immune biomarkers relevant to ART-treated HIV+ patients to facilitate future large-scale studies investigating individual differences in soy isoflavone metabolism within this patient population. Specifically, the short-term dose confirmation study will include those participants who are screened and meet eligibility which will be determined using results from a 12 hr fasting lipid panel which includes total cholesterol (TC), low density lipoproteins (LDL), high density lipoproteins (HDL), and triglycerides; health history; and the 2013 American College of Cardiology/ American Heart Association (ACC/AHA) Guidelines cardiovascular risk calculator. Eligible participants will be enrolled and then instructed to follow a legume-free diet (avoid beans, soy beans, lentils, bean sprouts, and peanuts) for two weeks, abstain from other vitamins or dietary supplements, and follow the provided standardized multivitamin regimen. Participants will return to clinic for a fasting blood collection and submit a 24 hour urine collection at week 0. At the end of this visit, participants will be instructed to consume one packet (10 pieces) of soy pretzels twice daily and continue to follow the legume-free diet with the provided multivitamin regimen. Participants will return after 4 weeks to obtain a second month's supply of study agents. Subjects will return after a second 4 weeks for a fasting blood collection and to submit a completed 24 hr urine collection. The subsequent placebo controlled study will include the same criteria used for the earlier short-term study. Participants will be randomized to either a soy pretzel intervention (1 packet of pretzels twice/day: total 20 pieces delivering 24g soy protein and ~60mg isoflavones) or a wheat pretzel intervention (placebo, 1 packet of pretzels twice/day: total 20 pieces containing 0g soy protein and 0mg isoflavones) for 12 weeks before crossing over to the other pretzel intervention for a second 12 weeks. A two-week washout period involving a legume-free diet and standardized multivitamin regimen, similar to the short-term study, will precede each intervention period. Blood and 24-hour urine will be collected at the specified time points to evaluate the sustained effects of the soy pretzel intervention on biomarkers of cardiovascular risk, immune function, and metabolites of isoflavone intervention. This study addresses an innovative approach of utilizing a dietary soy snack food to reduce cardiac risk and to explore multiple drivers of immune activation in HIV disease (pro-inflammatory lipids, microbial translocation, and the cytokines they induce) increasing the likelihood that we will generate results that impact clinically relevant indices of HIV disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Females and males aged 18 years or older.
* ACC/AHA 2013 Guidelines 10 year risk between <15%
* HIV-1 infection as documented by any licensed ELISA (enzyme-linked immunosorbent assay) test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 ribonucleic acid (RNA), or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* Receiving any stable Department of Health and Human Services (DHHS) recommended or alternative antiretroviral regimen for at least the last 12 weeks prior to study entry.
* Cumulative duration of antiretrovirals for at least 12 months at study entry.
* Documentation of at least 2 consecutive HIV-1 RNA levels of ≤50 copies/mL using any standard commercially assay for at least 6 months prior to study entry. An isolated (non-consecutive) HIV RNA > 50 copies/mL (but less than 400 copies/mL) within the previous 12 months is permitted.
* Provides written informed consent and is capable of reading and comprehending the informed consent.
* Meet Karnofsky performance status ≥70.
* Have a body mass index (BMI) between 20-35 kg/m2.
* Have a fasting total cholesterol levels of ≥200mg/dL AND either LDL cholesterol level of 120 to 190mg/dL or a HDL ≤ 40 mg/dL
* Laboratory values obtained at screening:

  * ANC (absolute neutrophil count) >1000/mm3
  * Hemoglobin >11 g/dL
  * Platelets ≥100,000/mm3
  * Calculated creatinine clearance (CrCl) >60 mL/min, as estimated by the Cockcroft-Gault equation
  * ALT (alanine aminotransferase) <5 x ULN (upper limit of normal) or ALT <3 x ULN and total bilirubin <1.5 x ULN Note: If the potential subject is taking an atazanavir-containing regimen at the time of screening, total bilirubin ≤5 x ULN is acceptable.
  * Hgb A1c (Hemoglobin A1c) ≤6.5%
* Have no plans to alter antiretroviral therapy (including structured treatment interruptions), diet (beyond soy intervention) or exercise regimens during the course of the study.
* Agree to collect urine for 24 hours and have blood collected, at specified time points.
* Agree to abstain from use of herbal or dietary supplements during the 6 weeks for the short-term study or 28 weeks for the placebo-controlled study or any other supplements that might interact with dietary soy intervention.
* Agree to follow a daily vitamin and mineral supplement regimen for 6 weeks for the short-term study or 28 weeks for the placebo-controlled study.
* Agree to abstain from legume foods or products made from these ingredients which are known to be high in isoflavones for 6 weeks or 28 weeks:

Soy: Edamame, Miso, Soy cheese, Tofu, Tempeh, Protein bars, Soymilk, Natto, Soy meat substitutes Beans: Navy, Kidney, Green beans, Lima, Pinto, Black beans, Cannellini, and Chickpeas Peas: Green, Snow, Black-eyed Peanuts: Peanuts, Peanut butter (1 tablespoon/week permitted) Sprouts: Alfalfa, Clover, Mung bean, Soybean

Exclusion Criteria:

* Need (or anticipated need in the next 24 weeks) for lipid modification pharmacotherapy or hypolipidemics (e.g., statins or fibrates) or hypoglycemic therapy.
* A clinically important illness within 14 days prior to study entry not explicitly excluded by the protocol, a physical or psychiatric disability, or a laboratory abnormality that might place the subject at increased risk by being exposed to the medications in this study or which might confound the interpretation of this investigation.
* Chronic hepatitis B or C infection Note: Participants who have been treated for their hepatitis C and have achieved a sustained virologic response (SVR) of 12 may participate.
* Any active or chronic uncontrolled inflammatory condition.
* Diarrhea or vomiting of Grade ≥ 2 within 14 days prior to study entry.
* An active AIDS-defining opportunistic infection or disease (for the purpose of this study, a cluster of differentiation 4 (CD4) count <200 cells/mm3 in the absence of any other AIDS-defining indicator condition is not considered an AIDS-defining event).
* Inability to maintain adherence to study schedule or communicate with study personnel.
* Current alcohol or recreational drug use which in the investigator's opinion interferes with the subject's ability to comply with dosing schedule and protocol evaluations.
* Any change in the last 24 weeks in therapy with prescription omega-3 fatty acids (>2 gram/day of Lovaza®), fibrates, or prescription niacin. Therapy with OTC (over the counter) omega 3 fatty acids or with ≤ 2 g Lovaza® is allowed. Any statin therapy for longer than 14 days received in the last 24 weeks is exclusionary.
* Have had a full treatment course/regimen of antibiotics 6 months prior to start of study.
* Known sensitivity or allergy or intolerance to wheat, soy, or any of the ingredients found in pretzels (yeast, soy bean oil, palm oil, or diastase enzymes).
* Have had a malignancy of any kind or ongoing chemotherapy, radiation therapy, or other cancer-related treatment.
* Concurrent use of immunosuppressant medications, including but not limited to immunomodulating agents, steroids, and chronic anti-inflammatory agents.
* Active metabolic or digestive illness including malabsorptive disorders, diabetes mellitus (indicated by Hgb A1c of ≥6.8% or on exogenous insulin therapy), renal insufficiency, hepatic insufficiency, hyper- or hypothyroidism, or short bowel syndrome, have an active or a recent history of any condition that causes altered immunity, co-morbid cardiac, pulmonary, renal, neurologic, and endocrine.
* Known underlying myositis or muscle disease.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hypertension, or psychiatric illness/social situation that would limit compliance with study requirements.
* Lack of regular access to a household freezer (for pretzel storage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-06; Primary Completion 2023-10 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Serious and Non-Serious Adverse Events with Pretzel Intervention (Division of AIDS Adverse Event version 2.0) | 6 weeks or 28 weeks
  Number of participants having adverse events with daily consumption of pretzels.
Self-Reported Daily Diary to Assess Adherence of Dietary Intervention | 6 weeks or 28 weeks
  Number of participants reporting 80% adherence to pretzels will have quantifiable levels of isoflavone (naturally occurring compounds in soy) metabolites in urine during soy pretzel intervention.

SECONDARY OUTCOMES:
Evidence of Improved lipid parameters in Antiretroviral Therapy Treated HIV+ patients with soy pretzel intervention | baseline to 6 weeks or baseline to 28 weeks
  Number of participants with changes in lipid parameters before (baseline) and after (6 or 28 weeks) after soy pretzel intervention
Evidence of Improved Arterial Function in Antiretroviral Therapy-Treated HIV+ Patients after Soy Pretzel Intervention | baseline to 6 weeks or baseline to 28 weeks
  Number of participants with changes in arterial function before (baseline) and after (6 or 28 weeks) after soy pretzel intervention
Evidence of Improved Immunologic Function of Soy Pretzels in Antiretroviral Therapy-Treated HIV+ patients | 28 weeks
  Ex vivo measurement of plasma markers of immune activation, inflammation and phenotypic analyses of monocyte and lymphocyte subpopulations during the dietary intervention will be coupled with in vitro assays aimed at assessing the mechanism(s) related to the modulation of inflammation and immune activation by soy metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Funderburg, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No